CLINICAL TRIAL: NCT05366439
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled Study to Assess the Antiviral Activity and Safety of AT-752 in a Dengue Human Challenge Model
Brief Title: Study of AT-752 in Healthy Subjects in a Dengue Human Challenge Model
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to deprioritize the dengue program
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-02A-003
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-05

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — AT-752

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AT-752 (Experimental): AT-752 administered orally for 14 days
  Interventions: Drug: AT-752
- Placebo (Placebo Comparator): Matching placebo administered orally for 14 days
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: AT-752 — Parallel Assignment
  Arms: AT-752
Drug: Placebo Comparator — Parallel Assignment
  Arms: Placebo

SUMMARY:
This study will assess the safety and antiviral activity of AT-752 in healthy subjects in a Dengue Human Challenge Model

DETAILED DESCRIPTION:
A Phase 1, double-blind, randomized, placebo-controlled study to assess the antiviral activity and safety of AT-752 in a Dengue Human Challenge Model

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use protocol-specified methods of contraception
* Negative pregnancy test
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Abuse of drugs
* Other clinically significant medical conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Mean quantitative RNAemia (peak and duration and area under the plasma concentration versus time curve [AUC]) | Day 2 until 28 days post virus inoculation

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Syracuse, New York, United States